CLINICAL TRIAL: NCT02694705
Title: Assessment of Preoxygenation Strategies in the Prehospital Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Essex and Herts Air Ambulance (Other)
Responsible Party: Principal Investigator, Christopher Groombridge, Dr, Queen Mary University of London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: QMERC2015/69
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia; Hypoxia
Keywords: Oxygen Inhalation Therapy; Intubation; Emergency Medicine
MeSH Terms: conditions — Hypoxia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CPAP (Experimental): 3 minutes of preoxygenation with a portable ventilator providing Continuous Positive Airway Pressure (CPAP) at 5 cmH20 and an FiO2 of 100%.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP)
- BVM (Experimental): 3 minutes of preoxygenation with a bag-valve-mask (BVM) device and oxygen flow rate of 15 litres / minute.
  Interventions: Device: Bag-Valve-Mask (BVM)
- NRM (Experimental): 3 minutes of preoxygenation with a non-rebreather mask (NRM) device and oxygen flow rate of 15 litres / minute.
  Interventions: Device: Non-rebreather Mask (NRM)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — CPAP provided by a portable Draeger Oxylog® 3000 plus ventilator
  Arms: CPAP
Device: Bag-Valve-Mask (BVM) — Preoxygenation provided by BVM device, oxygen flow rate 15 l/min
  Arms: BVM
Device: Non-rebreather Mask (NRM) — Preoxygenation provided by NRM, oxygen flow rate 15 l/min
  Arms: NRM

SUMMARY:
Comparison of the preoxygenation efficacy of tidal volume breathing using three different preoxygenation techniques which are available to providers in the prehospital environment.

DETAILED DESCRIPTION:
Prospective randomised interventional study.

Healthy volunteers will be positioned supine and undergo preoxygenation by tidal volume breathing for 3 minutes using each technique in turn. The sequence of techniques for each volunteer will be randomised in advance. Investigators will be instructed to ensure a good mask seal throughout the testing period. At the end of a 3 minute preoxygenation period, after a brief breath hold, the volunteer will exhale into reservoir tubing, allowing the fractional expired oxygen concentration (FeO2) to be determined (primary outcome) using a calibrated gas analyser.

The techniques being assessed have been chosen from methods of preoxygenation commonly available to clinicians in the prehospital environment:

1. Continuous Positive Airway Pressure mode with fractional inspired oxygen concentration (FiO2) 100% using a portable ventilator.
2. Bag-valve-mask device (BVM) with 15 l/min oxygen flow.
3. Non-rebreather mask (NRM) device with 15 l/min oxygen flow.

Volunteers will also be asked to indicate the subjective ease of breathing for each technique (secondary outcome) using a visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers

Exclusion Criteria:

* Pregnancy
* Respiratory disease
* Bearded
* Facial abnormality
* Edentulous

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fractional Expired Oxygen Concentration | 3 minutes
  Measure of denitrogenation efficacy

SECONDARY OUTCOMES:
Ease of breathing assessment using a visual analogue scale | 3 minutes
  Visual analogue scale to assess subjective ease of breathing through each device

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Groombridge, MBBS, Principal Investigator — Queen Mary University of London
Locations (1):
- Essex & Herts Air Ambulance Trust, Earls Colne, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groombridge C, Chin CW, Hanrahan B, Holdgate A. Assessment of Common Preoxygenation Strategies Outside of the Operating Room Environment. Acad Emerg Med. 2016 Mar;23(3):342-6. doi: 10.1111/acem.12889. Epub 2016 Feb 17. PMID 26728311